CLINICAL TRIAL: NCT02583685
Title: Efficacy and Safety of Switching From Pegylated Interferon/Ribavirin (PR) to Direct-acting Antiviral Agents (DAAs) for Chinese With CHC Genotype 1b Infection (SWITCH-1)
Brief Title: Switching Regimen in Treating Cirrhotic HCV GT1b Subjects
Acronym: SWITCH-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_SWITCH-1
Record Dates: First submitted 2015-10-12; First posted 2015-10-22 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — peginterferon alfa-2a; Ribavirin; ledipasvir, sofosbuvir drug combination; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- PR4 + LDV/SOF + ASV 4 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA <25 IU/ml by week 2 will receive LDV/SOF + ASV for 4 weeks.
  Interventions: Drug: PR4 + LDV/SOF + ASV 4 wk
- PR4 + LDV/SOF + SMV 4 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA <25 IU/ml by week 2 will receive LDV/SOF + SMV for 4 weeks.
  Interventions: Drug: PR4 + LDV/SOF + SMV 4 wk
- PR4 + LDV/SOF + ASV 6 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA <25 IU/ml by week 4 will receive LDV/SOF + ASV for 6 weeks.
  Interventions: Drug: PR4 + LDV/SOF + ASV 6 wk
- PR4 + LDV/SOF + SMV 6 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA <25 IU/ml by week 4 will receive LDV/SOF + SMV for 6 weeks.
  Interventions: Drug: PR4 + LDV/SOF + SMV 6 wk
- PR4 + LDV/SOF + ASV 8 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA > 2 log drop but ≥25 IU/ml by week 4 will receive LDV/SOF + ASV for 8 weeks.
  Interventions: Drug: PR4 + LDV/SOF + ASV 8 wk
- PR4 + LDV/SOF + SMV 8 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA > 2 log drop but ≥25 IU/ml by week 4 will receive LDV/SOF + SMV for 8 weeks.
  Interventions: Drug: PR4 + LDV/SOF + SMV 8 wk
- PR4 + LDV/SOF + ASV 12 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA <2 log drop by week 4 will receive LDV/SOF + ASV for 12 weeks.
  Interventions: Drug: PR4 + LDV/SOF + ASV 12 wk
- PR4 + LDV/SOF + SMV 12 wk (Experimental): Participants treated with 4 weeks pegylated interferon and ribavirin and plasma HCV RNA <2 log drop by week 4 will receive LDV/SOF + SMV for 12 weeks.
  Interventions: Drug: PR4 + LDV/SOF + SMV 12 wk

INTERVENTIONS:
Drug: PR4 + LDV/SOF + ASV 4 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Asunaprevir (ASV) 200mg administered orally twice daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; Sunvepra®
  Arms: PR4 + LDV/SOF + ASV 4 wk
Drug: PR4 + LDV/SOF + SMV 4 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Simeprevir (SMV) 150 mg tablet orally once daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; OLYSIO®
  Arms: PR4 + LDV/SOF + SMV 4 wk
Drug: PR4 + LDV/SOF + ASV 6 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Asunaprevir (ASV) 200mg administered orally twice daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; Sunvepra®
  Arms: PR4 + LDV/SOF + ASV 6 wk
Drug: PR4 + LDV/SOF + SMV 6 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Simeprevir (SMV) 150 mg tablet orally once daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; OLYSIO®
  Arms: PR4 + LDV/SOF + SMV 6 wk
Drug: PR4 + LDV/SOF + ASV 8 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Asunaprevir (ASV) 200mg administered orally twice daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; Sunvepra®
  Arms: PR4 + LDV/SOF + ASV 8 wk
Drug: PR4 + LDV/SOF + SMV 8 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Simeprevir (SMV) 150 mg tablet orally once daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; OLYSIO®
  Arms: PR4 + LDV/SOF + SMV 8 wk
Drug: PR4 + LDV/SOF + ASV 12 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Asunaprevir (ASV) 200mg administered orally twice daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; Sunvepra®
  Arms: PR4 + LDV/SOF + ASV 12 wk
Drug: PR4 + LDV/SOF + SMV 12 wk — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection; Ribavirin (RBV) administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg); Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally once daily; Simeprevir (SMV) 150 mg tablet orally once daily.
  Other Names: Pegasys®; Copegus®; Harvoni®; OLYSIO®
  Arms: PR4 + LDV/SOF + SMV 12 wk

SUMMARY:
This is a prospective, randomized study to evaluate the efficacy and safety of switching treatment from Peg-interferon and Ribavirin to direct-acting antiviral agents in Chinese with CHC genotype 1b infection, who are interferon/ribavirin-intolerant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with chronic HCV GT1b infection;
* HCV RNA ≥ 10000 IU/mL at screening;
* Received 4 weeks pegylated interferon plus ribavirin (PR4) therapy and are intolerant to PR4;
* Cirrhosis determination; a liver biopsy may be required;
* Use of highly effective contraception methods if female of childbearing potential or sexually active male;

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner;
* HIV or HBV co-infection;
* Hematologic or biochemical parameters at Screening outside the protocol- specified requirements;
* Active or recent history (≤ 1 year) of drug or alcohol abuse;
* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks (SVR12) after discontinuation of therapy | Post treatment Week 12
  SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after last dose of study drug.
Proportion of participants with adverse events leading to permanent discontinuation of study drug(s) | Baseline up to Week 24

SECONDARY OUTCOMES:
Proportion of participants with unquantifiable HCV viral load at specified time points during and after treatment | Baseline up to Week 24
Treatment adherence | Baseline to Week 12
  To evaluate the proportion of patients adherent to therapy (both on-treatment adherence and treatment discontinuation)
Change in health related quality of life evaluated with questionnaires | Up to Posttreatment Week 24
  To evaluate the change in health-related quality of life during and after treatment with questionnaires
Change in mental health evaluated with questionnaires | Up to Posttreatment Week 24
  To evaluate the change in mental health during and after treatment with questionnaires
Liver disease progression | Up to 10 years
  Liver disease progression is a composite endpoint measured by laboratory parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, albumin, platelets, prothrombin time (PT) and α-fetoprotein) and observed or reported clinical signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, Principal Investigator — Humanity and Health GI and Liver Centre
Locations (2):
- China (2):
  - Liver Fibrosis Diagnosis and Treatment Centre, 302 Hospital, Beijing, Beijing Municipality
  - Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong